CLINICAL TRIAL: NCT03868306
Title: Red Cell Distribution Width Index Versus Red Cell Distribution Width as Discriminating Guide for Iron Deficiency Anaemia and Beta Thalassemia Trait .
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rania, Principal investigator, Assiut University
Other Study IDs: RCDWIVRCDWADGFIDAABTT
Record Dates: First submitted 2019-03-07; First posted 2019-03-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Microcytic Hypochromic Anemia
MeSH Terms: conditions — Anemia, hypochromic microcytic | interventions — Blood Cell Count; Blood Protein Electrophoresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Iron deficiency anaemia: Microcytic hypochromic anaemic patients with serum ferritin less than 12 Ng /ml
  Interventions: Other: CBC , Iron study and Haemoglobin electrophoresis .
- Beta thalassemia Trait: Microcytic hypochromic anaemic patients with HBA2 more than 3.2 %
  Interventions: Other: CBC , Iron study and Haemoglobin electrophoresis .

INTERVENTIONS:
Other: CBC , Iron study and Haemoglobin electrophoresis . — The study will conducting on 100 patients of microcytic hypochromic anaemia who recruited from the hematology outpatient clinic , Assiut University Children Hospital . Beside history and clinical examination , the studied cases will be subjected to the following investigations Complete blood count ( CBC ) with comparison of MCV , RBCs count , RDW and RDWI . Determination of serum ferritin , serum iron and total iron bending capacity ( TIBC ) . HB electrophoresis . Patient with HBA2 more than 3.2 % are identified as beta thalassemia trait and patients with serum ferritin less than 12 ng / ml are identified as IDA cases. Validity of both discrimination indices are evaluated by calculating there sensitivity , specificity , positive predictive value , negative predictive value and Youden index ( YI ) Based on statistical criteria in ideal test should have high sensitivity and specificity and Youden index.

SUMMARY:
Red Cell Distribution Width Index versus Red Cell Distribution Width as Discriminating Guide for Iron Deficiency Anaemia and Beta Thalassemia Trait .

DETAILED DESCRIPTION:
Microcytic hypochromic anaemia is very common hematological abnormality in the clinical practice ( Snakar et;al. 2016 ) . Iron deficiency anaemia and beta thalassemia trait are the most common causes of microcytic hypochromic anaemia. As mentioned by the World Health Organization ( WHO ) estimates in 2004 , there were 273000deaths due to iron deficiency anaemia along with 19.7 million disability . Approximately 1.3 % cases were recorded globally in developing countries ( Kasseban et;al.2014 ) . Iron deficiency anemia is the most common nutritional disorder . This type of anemia is the final phase of a process that begins with exhaustion of iron stores and continues with iron depletion from other compartments that contain it compromising normal haematopoesis ( Wharton et;al. 1994 ) Beta thalassemia trait is the second most common cause of microcytic hypochromic anaemia . It is genetically determined disorder in which the defect of b globin gene results in decreased production of hemoglobin A1 ( Sliman et;al. 2004 ) The differentiation between Iron deficiency anemia and Beta thalassemia trait is important because of two main reasons . First , because hemoglobin will not improve in beta thalassemia trait if it is misdiagnosed as Iron deficiency anemia and unnecessary iron being prescribed by the attending physician ( Vehapoglee et;al. 2014 ) . The second grave reason is that misdiagnosed beta thalassemia trait as Iron deficiency anemia may get married to a beta thalassemia trait , resulting in homozygous or thalassemia major in the offsprings ( Tripathi et;al. 2015) Ideally one needs a battery of tests including detailed peripheral blood picture , HBA2 estimation , serum iron , TIBC , serum ferritin and transferrin saturation to differentiate Iron deficiency anemia from beta thalassemia trait clearly (Bordbar et;al. 2015 ) . But all these investigations are either not available in all clinical setup or they are relatively time consuming and need expensive techniques ( Natios et;al. 2007 ). Derived indices showed that RDW is the first index of the routine blood count to become abnormal during the development of Iron deficiency anemia ( McCulre et;al. 1985 ) . It quantitatively measures red blood cells size.

variation computed directly from the RBCs histogram and is calculated as standard statistical value , the coefficient of variation of the volume distribution ( Verma et;al. 2015 and Plengsures et;al. 2015) . RDW is high in Iron deficiency anemia because there is a wide variation in red cell size . in beta thalassemia trait , the red cells are all the same size , there is virtually no variation ,so RDW is low ( Park et;al.2009 ) . Another red cell discriminate function , RDWI had been proven to be reliable discrimination index in the differentiation between Iron deficiency anemia and beta thalassemia trait ( Ismail et;al.2016 ) . It can be easily calculated as ( MCV in ( Fl) x RDW / RBCs in (million per microlitre ) ) quotient more than 220 suggest Iron deficiency anemia

, less than 220 suggest beta thalassemia trait. RDWI provide valiable help to the attending physician as all discriminating factors including RBCs count , MCV and RDW are incorporated in its formula ( Jayabose et;al. 1999 ) .

ELIGIBILITY:
Inclusion Criteria:

* All patients with microcytic hypochromic anemia ( according to WHO , MCV less than 80 fl and HB level below the lower limit of normal value specified by age and gender .

Exclusion Criteria:

* Beta thalassemia major patients .
* Chronic diseases or infections .
* Lead poisoning .
* Sideroblastic anaemia .

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will conducting on 100 patients of microcytic hypochromic anaemia who recruited from the hematology outpatient clinic , Assiut University Children Hospital .
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic comparison of both the RDWI and RDW in the differentiation of Iron deficiency anemia and Beta thalassemia trait | Baseline
  RDW is high in Iron deficiency anemia because there is a wide variation in red cell size . in beta thalassemia trait , the red cells are all the same size , there is virtually no variation ,so RDW is low ( Park et;al.2009 ) . Another red cell discriminate function , RDWI had been proven to be reliable discrimination index in the differentiation between Iron deficiency anemia and beta thalassemia trait ( Ismail et;al.2016 ) . It can be easily calculated as ( MCV in ( Fl) x RDW / RBCs in (million per microlitre ) ) quotient more than 220 suggest Iron deficiency anemia
  , less than 220 suggest beta thalassemia trait.

IPD SHARING:
Plan to Share IPD: Undecided